CLINICAL TRIAL: NCT03800589
Title: Comparison of ExPress Implantation Versus Partial Deep Sclerectomy Combined With ExPress Implantation With Simultaneously Phacoemulsification
Brief Title: Assessment of Effectiveness Ex-Press Surgery Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/WIM/2010
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Glaucoma, Open-Angle; Glaucoma Secondary; Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Prospective, randomized control study with 24-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phaco and Ex-Press (Active Comparator): patients with co-existing cataract and glaucoma, qualified to the combined glaucoma surgery according to the protocol which were randomized to phacoemulsification with implantation of the Ex-Press
  Interventions: Procedure: phacoemulsification with implantation of the Ex-Press
- deep sclerectomy, phaco and Ex-press (Active Comparator): patients with co-existing cataract and glaucoma, qualified to the combined glaucoma surgery according to the protocol which were randomized to deep sclerectomy, phacoemulsification, ExPress implantation
  Interventions: Procedure: deep sclerectomy, phacoemulsification, ExPress implantation

INTERVENTIONS:
Procedure: phacoemulsification with implantation of the Ex-Press — The conjunctiva is dissected with the base in the limbus. A square scleral flap is dissected with the based in the limbus. Phacoemulsification is performed through a corneal incision 2.75 mm from the temple using the phaco-chop technique. Mini seton was implanted at 12 o'clock according to the standard technique.
  Arms: phaco and Ex-Press
Procedure: deep sclerectomy, phacoemulsification, ExPress implantation — The conjunctiva is dissected with the base in the limbus. Superficial flap is dissected with the based in the limbus. Phacoemulsification is performed through a corneal incision 2.75 mm from the temple using the phaco-chop technique. Deep scleral is dissected just below the trabeculo-Descemet membrane. The seton is implanted in the anterior chamber at the height of Schlemm's Canal.
  Arms: deep sclerectomy, phaco and Ex-press

SUMMARY:
The purpose of the study is to compare the effectiveness and safety profile of ExPress implantation versus partial deep sclerectomy combined with ExPress implantation with simultaneously phacoemulsification.

DETAILED DESCRIPTION:
Mermoud et all (1) proposed a modification of the classical surgical technique: combined deep sclerectomy (DS) with ExPress device implantation. The goal of this modification was to enhance hypotensive effect of well known procedure, and also to simplify non-penetrating surgery, which is a procedure with a long learning curve. Mermoud's idea provides the possibility of avoiding complications related to dissection of the filtering bleb and gives hope for achieve of better results in comparison to the classical procedure. Thanks to this, the surgical procedure could be performed earlier, even in the case of glaucoma with low intraocular pressure (IOP), where vascular factors are largely responsible for the progression of neuropathy. To demonstrate the potential of both types of procedures with the application of the ExPress implant, the authors decided to conduct a prospective, randomized study with a 2-year observation period concerning the efficacy, safety and stability of effects achieved.

ELIGIBILITY:
Inclusion Criteria:

* co-existing glaucoma and cataract (NC1, NC2) classified by means of the LOCS III scale
* patients with primary open-angle glaucoma (POAG), pseudoexfoliative glaucoma (PGX) and normal tension glaucoma (NTG), in which a satisfactory IOP level was not achieved despite maximum tolerable hypotensive treatment, both topical and systemic,
* documented progression of loss of field of vision,
* significant daily IOP fluctuations,
* no cooperation from patient with regard to application of anti-glaucoma treatment,
* allergy to topical medication
* written consent to involvement and participation in the study for a period of at least 24 months

Exclusion Criteria:

* no consent to participation in the study
* prior surgical and laser procedures in the area of the eye
* narrow- or closed-angle glaucoma
* post-inflammatory or post-traumatic secondary glaucoma
* chronic illness of the cornea or optic nerve
* advanced macular degeneration
* active inflammatory process
* pregnancy
* systemic steroid therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
IOP | baseline, and 24th month after surgery
  the change in level of intraocular pressure
CDVA | baseline, and 24th month after surgery
  the change in corrected distance visual acuity
number of drugs | baseline, and 24th month after surgery
  the change in number of antiglaucoma medications

SECONDARY OUTCOMES:
number of complications | in a day of surgery
  rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Marek Rękas, Prof, Principal Investigator — Military Institute of Medicine in Warsaw

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 18 months of study completion
Access Criteria: Data access requests will be reviewed by the Chair Person. Requestors will be required to sign a Data Access Agreement

REFERENCES:
- [Result] Bissig A, Feusier M, Mermoud A, Roy S. Deep sclerectomy with the Ex-PRESS X-200 implant for the surgical treatment of glaucoma. Int Ophthalmol. 2010 Dec;30(6):661-8. doi: 10.1007/s10792-010-9382-z. Epub 2010 Jun 16. PMID 20552258